CLINICAL TRIAL: NCT03560037
Title: Use of Endocuff Vision to Increase Detection of Sessile Serrated Adenomas During Screening Colonoscopy
Brief Title: Use of a Distal Colonoscope Attachment to Increase Detection of Sessile Serrated Adenomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1164295
Record Dates: First submitted 2018-04-10; First posted 2018-06-18 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sessile Serrated Adenoma

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled to receive either conventional colonoscopy or colonoscopy with addition of Endocuff Vision device.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Colonoscopy (No Intervention): Patients randomly assigned to this group will receive standard colonoscopy without the use of a distal attachment.
- Endocuff Vision Assisted Colonoscopy (Experimental): Patients randomly assigned to this group will receive colonoscopy with the use of the Endocuff Vision distal attachment.
  Interventions: Device: Endocuff Vision Assisted Colonoscopy

INTERVENTIONS:
Device: Endocuff Vision Assisted Colonoscopy — Detachable device that is fixed to the end of colonoscope. The device has single-row of soft, hair-like projections that flatten colonic folds during colonoscope withdrawal which can aid in detection of colon polyps.
  Arms: Endocuff Vision Assisted Colonoscopy

SUMMARY:
This study evaluates whether the use of a disposable colonoscope attachment, Endocuff Vision, can increase the detection of sessile serrated adenomas. Participating patients will be randomized to receive either standard colonoscopy or colonoscopy with the Endocuff Vision.

DETAILED DESCRIPTION:
Colon cancer remains the second leading cause of death amongst both men and women in the United States(1). With the advent of screening colonoscopy, mortality from colorectal cancer has decreased, and colonoscopy is the current gold standard for colorectal cancer screening and prevention by removing adenomatous polyps.

Different devices have been employed to assist the endoscopist in the detection of colon adenomas, as these lesions serve as precursors to colon neoplasia. One device of interest is the Endocuff Vision. The Endocuff Vision is a disposable device with a single row of soft, hair-like projections that aid in flattening colonic folds during colonoscope withdrawal to increase the detection of colon adenomas. Previous studies have compared endocuff-assisted colonoscopy to standard colonoscopy, and the results have indicated significant improvement in overall adenoma detection rates (ADR)(2-4). All of these studies have focused on the detection of conventional tubular adenomas as primary endpoints. However, there exists an additional serrated adenoma pathway that may give rise to about 15-20% of colon cancers (5). These lesions tend to be flatter with subtler features that make them harder to detect. A recent meta-analysis suggested that the endocuff was more effective at detecting sessile serrated adenomas compared to standard colonoscopy; however, these findings are derived from secondary data analyses (6). To the best of our knowledge, no study to date has examined the sessile serrated adenoma detection rate as a primary endpoint.

Our previous study examined the differences in overall adenoma detection between endocuff-assisted and standard colonoscopy. Although there was no statistical difference in ADR between endocuff-assisted colonoscopy and standard colonoscopy, investigators did observe a numeric difference in sessile serrated adenoma detection rate (SSADR), 16.7% vs 23.8% (p = 0.5) between standard colonoscopy and endocuff-assisted colonoscopy, respectively. Given the previous sample size was calculated to detect differences in overall ADR, the study was not powered to determine whether this observed difference in SSADR was significant.

Therefore, the goal of the proposed study is to compare standard colonoscopy to endocuff-assisted colonoscopy in patients undergoing colonoscopy for colon cancer screening to determine differences in sessile serrated adenoma detection rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to our outpatient gastroenterology suites for screening colonoscopy.

Exclusion Criteria:

* Age less than 45 and greater than 85
* Prior history of colon polyps (hyperplastic polyp, tubular adenoma or sessile serrated adenoma) and colon cancer
* Patients with inflammatory bowel disease
* Patients suspected to have colon cancer based on non-invasive tests such as stool tests for hemoglobin or DNA, or imaging finding suggestive of colon cancer (CT or barium enema).
* Patients undergoing colonoscopy for evaluation of symptoms such as abdominal pain, rectal bleeding, diarrhea, constipation, etc., or patient with iron deficiency anemia suspected to be due to ongoing bleeding inside the colon
* Patients with family history of colon cancer in 1st degree relative below the age of 60
* Patients with family history of hereditary polyposis syndromes such as Lynch syndrome, familial adenomatous polyposis etc., which are associated with an increased risk of colon cancer
* Patients unable to consent
* Pregnant patients
* Incarcerated patients

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All patient de-identified data that is collected during the clinical trial.
Supporting Information: Study Protocol
Time Frame: Immediately after publication and ending at 5 years after publication.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Background] De Palma GD, Giglio MC, Bruzzese D, Gennarelli N, Maione F, Siciliano S, Manzo B, Cassese G, Luglio G. Cap cuff-assisted colonoscopy versus standard colonoscopy for adenoma detection: a randomized back-to-back study. Gastrointest Endosc. 2018 Jan;87(1):232-240. doi: 10.1016/j.gie.2016.12.027. Epub 2017 Jan 9. PMID 28082115
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] Obuch JC, Ahnen DJ. Colorectal Cancer: Genetics is Changing Everything. Gastroenterol Clin North Am. 2016 Sep;45(3):459-76. doi: 10.1016/j.gtc.2016.04.005. PMID 27546843
- [Background] Chin M, Karnes W, Jamal MM, Lee JG, Lee R, Samarasena J, Bechtold ML, Nguyen DL. Use of the Endocuff during routine colonoscopy examination improves adenoma detection: A meta-analysis. World J Gastroenterol. 2016 Nov 21;22(43):9642-9649. doi: 10.3748/wjg.v22.i43.9642. PMID 27920485

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Started | 216 | 211
Completed | 215 | 210
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy | Total
Number analyzed (Participants) | 216 | 211 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (7.2) | 57.9 (7.7) | 57.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 92 | 206
  Male | 102 | 119 | 221
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.7 (4.9) | 27.6 (4.6) | 27.7 (4.8)
Alcohol consumption [Count of Participants; unit: Participants] — Yes or No
  Participants
    Yes | 153 | 145 | 298
    No | 63 | 66 | 129
Smoking [Count of Participants; unit: Participants] — Never/Former/Current Smoking
  Participants
    Never | 151 | 155 | 306
    Former | 55 | 50 | 105
    Current | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Sessile Serrated Adenomas
Description: Number of colonoscopies with at least one sessile serrated adenoma
Time Frame: Time point of assessment will be when pathology results are made available 2 weeks after procedure. Data will be collected through study completion, analyzed and reported up to 6 months after study completion.
Population: Participants with complete colonoscopy
Measure: Number; unit: colonoscopies
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
colonoscopies | 42 | 59

2. Secondary Outcome: Adenoma Detection
Description: Number of colonoscopies with at least one adenoma
Time Frame: as for outcome 1
Population: Participants with complete colonoscopy
Measure: Number; unit: colonoscopies
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
colonoscopies | 159 | 199

3. Secondary Outcome: Proximal Colon Adenomas
Description: Number of colonoscopies with at least one sessile serrated adenoma or conventional adenoma
Time Frame: as for outcome 1
Measure: Number; unit: colonoscopies
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
colonoscopies | 83 | 99

4. Secondary Outcome: Adenomas Per Colonoscopy
Description: Total adenomas detected in each treatment arm divided amongst the number of patients in each arm
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: adenomas per participant
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
adenomas per participant | 0.96 (1.33) | 1.24 (1.67)

5. Secondary Outcome: Sessile Serrated Adenomas Per Colonoscopy
Description: Total sessile serrated adenomas in each treatment arm divided amongst the number of patients in each arm.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sessile Serrated Adenomas Per Participan
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
Sessile Serrated Adenomas Per Participan | 0.27 (0.59) | 0.35 (0.74)

6. Secondary Outcome: Adenomas Per Positive Colonoscopy
Description: The total adenomas detected divided by the number of colonoscopies with at least one adenoma
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Adenomas Per Positive Colonoscopy
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
Adenomas Per Positive Colonoscopy | 1.97 (1.27) | 2.12 (1.71)

7. Secondary Outcome: Sessile Serrated Adenomas (SSA) Per Positive Colonoscopy
Description: The total sessile serrated adenomas detected divided by the number of colonoscopies with at least one sessile serrated adenoma
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: SSA Per Positive Colonoscopy
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
SSA Per Positive Colonoscopy | 1.20 (0.63) | 1.48 (0.82)

8. Secondary Outcome: Colonoscope Withdrawal Time
Description: The time it takes to withdraw the colonoscope from the cecum to the end of the examination.
Time Frame: Time point of assessment will be recorded at the time of colonoscopy. This data will be collected through study completion, analyzed and reported up to 6 months after study completion.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
minutes | 14.74 (0.28) | 15.01 (0.31)

9. Secondary Outcome: Differences in Quality of Bowel Preparation
Description: Measurement of colon preparation based on the validated Boston Bowel Prep Score. Each colon segment (right, transverse, and left colons) will receive a score of 0 (worse) to 3 (best). The sum of each segment will be reported as a total score of 0 (worse) to 9 (best).
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale (0 to 9)
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
Number analyzed (Participants) | 215 | 210
score on a scale (0 to 9) | 8.7 (0.8) | 8.7 (0.9)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Standard Colonoscopy | Endocuff Vision Assisted Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/211
Other Adverse Events (participants affected / at risk) | 0/216 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03560037/Prot_000.pdf
  • Informed Consent Form (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT03560037/ICF_001.pdf